CLINICAL TRIAL: NCT00231179
Title: The MOM Program Continuation - 5 Year Follow-up
Brief Title: The MOM Program: 5 Year Follow-up Study of a Home Visiting Program at The Children's Hospital of Philadelphia
Acronym: MOM Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: William Penn Foundation (Other); Claneil Foundation, Inc. (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2003-10-3495
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Child Development
Keywords: child, preschool; intelligence; environment; home visiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home visiting Intervention (Experimental): Home visiting intervention group.
  Interventions: Behavioral: Home visiting professional support model
- Control (Placebo Comparator): Control condition did not receive any services.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Home visiting professional support model — Home visits and telephone calls keyed to well child visits.
  Arms: Home visiting Intervention
Other: Control — The control group received an information booklet on child/family services upon enrollment and transportation for the follow-up evaluations. They were called every 4 months to maintain contact information
  Other Names: No intervention, informational booklet only
  Arms: Control

SUMMARY:
The purpose of the MOM Program Continuation is to promote child development by helping families become more competent in accessing and using available health, developmental and educational resources. The program focuses are childhood immunizations, Early Intervention services, lead screening, Early Head Start and Head Start enrollment. The Intervention consists of frequent phone calls and home visits to encourage mothers to have their babies immunized on schedule and to participate in needed developmental and educational services. The program seeks to fill the gap between children's need for services and mothers' ability to assure their children's participation in those services.

DETAILED DESCRIPTION:
The MOM Program Continuation builds on the work of The MOM Program, a 3 year randomized intervention. The premise of the MOM Program was that professional support through home visits and frequent phone contacts would improve children's cognitive and behavioral development, ultimately improving their early educational success. The children were enrolled in the MOM Program at birth. The MOM Program Continuation provides continued intervention for the children and mothers of the original cohort to assure that the children are prepared for kindergarten entry at 5 years of age and to evaluate the children's cognitive and behavioral outcomes at age 5 years. The program will also create a longitudinal database to study the linkages between maternal cognitive ability and child cognitive, educational, and behavioral outcomes through entry into school.

ELIGIBILITY:
Inclusion Criteria: Previous enrollment in The MOM Program; child age of 5 years (plus or minus 3 months); willingness to come to office for follow-up assessment visit; parental consent and child assent.

Exclusion Criteria: None.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2004-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerilynn Radcliffe, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Hospital of the University of Pennsylvania after giving birth to a healthy singleton newborn infant, if they lived in pre-identified ZIP Code areas of Philadelphia. Participants were recruited from July 6, 2001 through January 7, 2002. 302 mothers were enrolled and 254 completed the 5-year follow-up visit.
Pre-assignment Details: Randomization occurred at enrollment. At the time of follow-up, participants continued to remain in the originally assigned group of either control or intervention.
Groups:
- Home Visiting Intervention: The intervention group received home visits and follow up calls keyed to well child visits following American Academy of Pediatric guidelines. Follow-up and reminder calls were made to track health care visits completed and referrals made.
Period: Overall Study
Arm/Group | Home Visiting Intervention | Control
Started | 152 | 150
Completed | 128 (128 (95%) in intervention group completed the five year follow-up visit.) | 126 (126 (93%) in the control group completed the five year follow-up visit.)
Not Completed | 24 | 24
Not completed — Lost to Follow-up | 21 | 21
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Visiting Intervention | Control | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Customized [Number; unit: participants]
  4-5 years | 152 | 150 | 302
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 82 | 163
  Male | 71 | 68 | 139
Region of Enrollment [Number; unit: participants]
  United States | 152 | 150 | 302

OUTCOME MEASURES:

1. Primary Outcome: Wechsler Preschool and Primary Scale of Intelligence, Third Edition (WPPSI-III)
Description: Cognitive ability was assessed through the Wechsler Preschool and Primary Scale of Intelligence, Third Edition (WPPSI-III). The WPPSI-III has been developed and standardized for children ages 2 years, 6 months through 7 years, 3 months of age. The WPPSI-III yields a Verbal Score, a Performance Score, a General Language Score, and a Full Scale Score. These scores have a mean of 100 and a standard deviation of 15. The range of possible values is 50 (worst value) to 150 (best value).
Time Frame: 5 years of age (plus or minus 1 month)
Population: Number of children evaluated at 60 month visit.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Home Visiting Intervention | Control
Number analyzed (Participants) | 128 | 126
Scores on a scale | 86.5 (12.6) | 87.4 (12.2)
Statistical Analysis 1: Comparison: Home Visiting Intervention vs Control; We compared scores for verbal, performance, and full scale Intelligence Quotient (IQ); Test type: Non-Inferiority or Equivalence — Sample sizes were established when the trial was first developed. For all power calculations, we set alpha = .05 and beta = .20 and specified 2-tailed tests; p = 0.59, t-test, 2 sided — Bonferroni corrections were made for multiple comparisons; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [0.31 to 2.13], Standard Deviation 15.0

2. Primary Outcome: Child Behavior Checklist Internalizing Scale at 5 Years of Age, Percentage of Participants
Description: Caregivers completed The Child Behavior Checklist (CBCL) Preschool form from The Achenbach System of Empirically Based Assessment (ASEBA). The CBCL is standardized for children ages 1.5 to 5 years and measures child internalizing and externalizing behaviors and total problems. Respondents are asked to rate 99 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child" based on the past two months. The range of possible values is 0-100. Percentage of Participants with Abnormal Behavior is calculated by: % abnormal = # of Abnormal / (# of Normal + # of abnormal).
Time Frame: at child age of 5 years (plus or minus 1 month)
Population: Number of mothers/caregivers evaluated at 60 month visit.
Measure: Number; unit: percentage of participants
Arm/Group | Home Visiting Intervention | Control
Number analyzed (Participants) | 128 | 126
percentage of participants | 8 (8.9) | 11 (11.2)
Statistical Analysis 1: Comparison: Home Visiting Intervention vs Control; Test type: Non-Inferiority or Equivalence — Please see earlier power calculation; p = 0.72, Chi-squared; Hazard Ratio (HR) = 10, Standard Error of Mean 5

3. Primary Outcome: Child Behavior Checklist Externalizing Scale, Percentage of Abnormality in Participants
Description: as for outcome 2
Time Frame: at child age of 5 years (plus or minus 1 month)
Measure: Number; unit: percentage of participants
Arm/Group | Home Visiting Intervention | Control
Number analyzed (Participants) | 128 | 126
percentage of participants | 3 | 12
Statistical Analysis 1: Comparison: Home Visiting Intervention vs Control; Test type: Non-Inferiority or Equivalence — See previous; p < 0.01, Chi-squared; Hazard Ratio (HR) = 10, Standard Error of Mean 5

4. Primary Outcome: Child Behavior Checklist Aggressive Subscale, Percentage of Abnormality in Participants
Description: as for outcome 2
Time Frame: at child age of 5 years (plus or minus 1 month)
Measure: Number; unit: Percentage of participants
Arm/Group | Home Visiting Intervention | Control
Number analyzed (Participants) | 128 | 126
Percentage of participants | 4 | 12
Statistical Analysis 1: Comparison: Home Visiting Intervention vs Control; Test type: Non-Inferiority or Equivalence — See previous; p < 0.05, Chi-squared; Hazard Ratio (HR) = 3, Standard Error of Mean 3

5. Primary Outcome: Child Behavior Checklist Attention Subscale, Percentage of Abnormality in Participants
Description: as for outcome 2
Time Frame: child age 5 years (plus or minus 1 month)
Measure: Number; unit: Percentage of participants
Arm/Group | Home Visiting Intervention | Control
Number analyzed (Participants) | 128 | 126
Percentage of participants | 7 | 8
Statistical Analysis 1: Comparison: Home Visiting Intervention vs Control; Test type: Non-Inferiority or Equivalence — See previous; p = 0.64, Chi-squared; Hazard Ratio (HR) = 3, Standard Error of Mean 3

ADVERSE EVENTS:
Arm/Group | Home Visiting Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/150
Other Adverse Events (participants affected / at risk) | 0/152 | 0/150

LIMITATIONS AND CAVEATS:
The initial high rate of refusal to participate in the study may affect the generalizability of our results. Those who refused study participation were older and did not elaborate on their lack of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No